CLINICAL TRIAL: NCT05482815
Title: Evaluation of the Safety and Efficacy of Voice Prosthesis in Voice Reconstruction After Total Laryngectomy: a Prospective, Multicenter, Self-controlled Clinical Trial
Brief Title: Evaluation of the Safety and Efficacy of Voice Prosthesis in Voice Reconstruction After Total Laryngectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Atos Medical AB (Industry)
Collaborators: Peking Union Medical College Hospital (Other); Beijing Tongren Hospital (Other); Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMAB-FYN-1.0
Record Dates: First submitted 2022-07-26; First posted 2022-08-01 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Laryngectomy; Status
Keywords: Voice rehabilitation

STUDY DESIGN:
Intervention Model Description: prospective, multicenter, single-group test target trial design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Voice Prosthesis (Experimental): Subjects receive a Voice prosthesis using the Provox Puncture Set, then undergo an articulation training program (3 weeks). The voice prosthesis is replaced after 3 months and 6 months.
  Interventions: Device: Provox Vega Voice prosthesis

INTERVENTIONS:
Device: Provox Vega Voice prosthesis — Voice prosthesis for speech rehabilitation, Provox Vega Voice prosthesis

SUMMARY:
The objective of the study is to evaluate the clinical safety and efficacy of voice prosthesis for voice reconstruction after total laryngectomy in China.

Main outcome will be the assessment of pronunciation effect (subjective auditory assessment).

ELIGIBILITY:
Inclusion Criteria:

* The age is greater than 18 years; the gender is not limited
* Performed total laryngectomy;
* No voice prosthesis has been installed
* Be able to take care of themselves mentally and physically, and have good hand coordination ability
* With healthy wall sharing with trachea and esophagus
* The patient has a desire to restore articulation function
* Can speak Mandarin and have a certain reading ability (equivalent to primary school education)
* The subject is fully aware of the benefits and risks of this trial and is willing to participate in and sign the informed consent form

Exclusion Criteria:

* There is serious respiratory system disease or defect
* There is a serious skin disease in the tracheostoma
* Obvious intelligence and mental disorder
* Tracheostoma is narrow and needs cannula implantation
* Patients with limitation of mouth opening and other subjects with dyslalia or language disorders (such as subjects with sequelae of cerebral infarction, etc.)
* Patients with severe respiratory disease, cardiopulmonary disease (e.g., severe arrhythmia, persons with slow ventricular rate (ventricular rate <50 beats/ min), acute phase of myocardial infarction and severe heart failure), disturbances of blood coagulation (coagulation index PT, APTT, INR> 1.5 times of the normal upper limit), septicemia and other patients not suitable
* Patients with severe diseases of liver and renal function (liver function index, alanine aminotransferase (ALT), aspartate aminotransferase (AST)> 2 times of normal upper limit, renal function index, urine creatinine (Cr), blood urea nitrogen (BUN)> 2 times of normal upper limit);
* Patients with local recurrence of tumor or metastatic tumor
* If the patient has received esophageal articulation training, the time of training and using esophagus to speech should be less than 6 months
* Women planning to have child, in lactation or pregnancy during the whole clinical study
* Participated in other clinical trials within 1 month
* Other candidates the investigators think not appropriate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in pronunciation effect (subjective auditory assessment) | Baseline, 3 months, 6 months
  Voice recordings judged by two independent evaluators, scored from 1-7, with lower scores meaning worse speech.

SECONDARY OUTCOMES:
Change in longest articulation time (continuous /a/, count) | Baseline, 3 months, 6 months
  The longest duration time of one continuous / a / is recorded by a stopwatch, count and the average of three times are taken at the same time.
Change in sound intensity (minimum / maximum / comfortable); | Baseline, 3 months, 6 months
  Sound intensity of the minimum / maximum / comfortable loudness (measured 3 times per person) is recorded to calculate the dynamic range (in decibels)
Change in total time required to read a text | Baseline, 3 months, 6 months
  Standard Chinese text is read out loud, and the total time is recorded.
Change in Voice Handicap Index | Baseline, 3 months, 6 months
  Validated tool to assess Voice handicap. Statements on participant's voice quality and effect on social life are assessed by a five-point Likert-scale, ranged from 0-4, with high scores indicating more handicap (0 = Never, 4 = Always).
Change in Quality of Life by SF-36 | Baseline, 3 months, 6 months
  Patient reported, 36-item, Score of calculated, ranging from 0-100, the lower the score the more disability. The higher the score the less disability
Evaluation of operative performance | Baseline, 3 months, 6 months
  Study-specific questionnaire on feasibility and satisfaction of clinicians
Incidence of Adverse Events | Baseline, 3 months, 6 months
  Any adverse events (including serious adverse events and device defect rates) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Gao Zhiqiang, Chief Physician, Principal Investigator — Peking Union Medical College Hospital
Locations (3):
- China (3):
  - Beijing Tongren Hospital, CMU, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Eye & ENT Hospital of Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No